CLINICAL TRIAL: NCT01160848
Title: A Clinical Study of Photoactive Porphyrins (PAP) Levels in Acne-affected Skin After Topical Visonac Application in Patients With Moderate to Severe Facial Acne Vulgaris
Brief Title: Photoactive Porphyrins (PAP) Levels After Topical Visonac Application in Acne Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PC TA205/10
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Acne Vulgaris
Keywords: Moderate to severe Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Saline Waters; Salicylic Acid; Ethanol; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Other): Three areas will be randomized to either a pre-treatment cleaning using a wipe containing an ethyl alcohol solution(one area) or a cleansing wipe containing saline water (two areas), before application of the Visonac cream. One of the areas cleaned with saline wipe will also be occluded with a transparent dressing (Tegaderm) during the incubation time. In vivo fluorescence spectroscopy will be performed in the three areas before cream application, and at 1h, 1.5h, 2h, 2.5h and 3 h after cream application
  Interventions: Drug: Area cleaned with saline water and occluded with Tegaderm; Drug: Area cleaned with saline water; Drug: Area cleaned with Ethyl alcohol solution
- Part 2 (Other): For each patient, 3 areas were randomized to treatment with Visonac for 24 hours (2 areas) or Visonac for 1 hour (1 area)
  Interventions: Drug: Visonac left on the skin for 24 hours in facial area one; Drug: Visonac wiped off after one hour; Drug: Visonac left on the skin 24 hours in facial area two

INTERVENTIONS:
Drug: Area cleaned with saline water and occluded with Tegaderm
  Arms: Part 1
Drug: Area cleaned with saline water
  Arms: Part 1
Drug: Area cleaned with Ethyl alcohol solution
  Arms: Part 1
Drug: Visonac left on the skin for 24 hours in facial area one
  Arms: Part 2
Drug: Visonac wiped off after one hour
  Arms: Part 2
Drug: Visonac left on the skin 24 hours in facial area two
  Arms: Part 2

SUMMARY:
Open, prospective, randomized, single-centre study in patients with moderate to severe facial acne vulgaris. Three circular areas with a diameter of 4 cm, each circle including at least 4 inflammatory lesions, will be selected in acne-affected areas in the face. One area should be identified on each cheek and one area should be identified on the forehead. The minimum distance between the three areas should be at least 4 cm. For each patient the three areas will be randomized to either a pre-treatment cleaning using a wipe containing an ethyl alcohol solution(one area) or a cleansing wipe containing saline water (two areas), before application of the Visonac cream. One of the areas cleaned with saline wipe will also be occluded with a transparent dressing (Tegaderm) during the incubation time. In vivo fluorescence spectroscopy will be performed in the three areas before cream application, and at 1h, 1.5h, 2h, 2.5h and 3 h after cream application. After the last fluorescence spectroscopy reading, the cream should be wiped off and the patient should protect the three areas from sunlight, prolonged, or intense light for 2 days.

The study was extended with additionally 8 patients to explore the photoactive porphyrin levels over a 24 hour period:

The patients will clean their face with Cetaphil Gentle Skin Cleanser before cream application. For each patient the three areas will be randomized to Visonac 80mg left on the skin for 24 hours and Visonac (MAL8%) to be wiped of after 1 hour.

In vivo fluorescence spectroscopy will be performed at all three areas before cream application, and at 2h, 3 h, 4h, 5h, 8h, 10h, 11h, 12h, 13h, 15 and 24h after cream application. The exact time points may be adjusted based on the result from the previously included patients. All patients will be instructed to protect the three areas from sunlight, prolonged, or intense light for 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed and verified informed consent form. For patients under age of 18, an assent form in conjunction with an informed consent form, signed and verified by parent/guardian.
* Adolescent and adult female and male patients, from 12 to 35 years of age.
* Patients with moderate to severe facial acne vulgaris according to the IGA scale.
* Female patients who are surgically sterile, pre-menstrual, postmenopausal, abstinent, or willing to use an adequate means of contraception including birth control pills, or barrier methods and spermicide for at least 14 days prior to the study visit.
* Patients with skin type II to III (Fitzpatrick).
* Patients with 3 areas of 4 cm in diameter, each including at least with at least 4 inflammatory lesions (papules, pustules, and nodules) in the face (at cheek and forehead).

Exclusion Criteria:

* Subject is the investigator or any sub investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Patients unlikely to comply with the protocol, e.g. mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the clinical study, uncooperative attitude or unlikelihood of completing the study (e.g. drug or alcohol abuse).
* Female subjects with childbearing potential (i.e. ovulation, pre-menopausal, not surgically sterilized) not willing to use a medically accepted contraceptive regimen while on treatment.
* Pregnancy
* Lactating.
* Participation in other clinical studies either currently or within the last 30 days.
* Patients with porphyria.
* Known allergy to (MAL), to a similar PDT compound, or to excipients of the cream
* Patients with cutaneous photosensitivity.
* Patients that have received topical treatments for their acne within the last 14 days. Medicated cleansers not containing active ingredients such as 5% BPO or high concentration of salicylic acid may be stopped before the treatment. (Cosmetic Cleansers that contains no more than 2 % salicylic acid is allowed).
* Patients that has received oral antibiotics for treatment of their acne within the last month.
* Patients that has received oral isotretinoin within the last 6 months.
* Patients with a beard that might interfere with study assessments.
* Patients with melanoma or dysplastic nevi in the treatment area

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael T. Jarratt, M.D., Principal Investigator — Derm Research, PLLC
Locations (1):
- DermResearch, Inc., Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in one center in the US:
  Michael Jarratt M.D. DermResearch Inc. 8140 N Mopac Building 3, Suite 120 Austin, TX 78759. First patient entered the study on the 8th of November 2010 Last patient last visit on the 9th January 2011
Groups:
- 3 Areas Per Patient, 3 Hours: Visonac : MAL 80 mg/g Group 1: Alcohol wipe and Visonac without occlusion Group 2: Saline wipe and Visonac with occlusion Group 3: Saline wipe and Visonac without occlusion
- 3 Areas Per Patient, 24 Hours: Group 1: Visonac left on skin for 1 hour Group 2: Visonac left on skin for 24 hours, area 1 Group 3: Visonac left on skin for 24 hours, area 2
Period: Overall Study
Arm/Group | 3 Areas Per Patient, 3 Hours | 3 Areas Per Patient, 24 Hours
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Areas Per Patient, 3 Hours | 3 Areas Per Patient, 24 Hours | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 8 | 15
  Between 18 and 65 years | 5 | 0 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20
Fluoresence intensity [Mean (Full Range); unit: Fluoresence intensity unit] — In the study arm "3 Areas Per Patient, 3 Hours", participants were only treated with "Alcohol wipe and Visonac without occlusion", "Saline wipe and Visonac with occlusion", "Saline wipe and Visonac without occlusion".
  In the study arm "3 Areas Per Patient, 24 Hours" participants were only treated with "Visonac left on skin for 1 hour", "Visonac left on skin for 24 hours, area 1", "Visonac left on skin for 24 hours, area 2".
  Fluoresence intensity unit
    Alcohol wipe and Visonac without occlusion | 10.5 (5.0) [4 to 17.5] | NA [NA to NA] — Participants in this study arm were not provided this treatment, please see Baseline Measure Description. | 10.5 [4 to 17.5]
    Saline wipe and Visonac with occlusion | 11.2 [5 to 28] | NA [NA to NA] — Participants in this study arm were not provided this treatment, please see Baseline Measure Description. | 11.2 [5 to 28]
    Saline wipe and Visonac without occlusion | 10.8 [5 to 17] | NA [NA to NA] — Participants in this study arm were not provided this treatment, please see Baseline Measure Description. | 10.8 [5 to 17]
    Visonac left on skin for 1 hour | NA [NA to NA] — Participants in this study arm were not provided this treatment, please see Baseline Measure Description. | 9.3 [3 to 20.5] | 9.3 [3 to 20.5]
    Visonac left on skin for 24 hours, area 1 | NA [NA to NA] — Participants in this study arm were not provided this treatment, please see Baseline Measure Description. | 10.5 [4 to 19.5] | 10.5 [4 to 19.5]
    Visonac left on skin for 24 hours, area 2 | NA [NA to NA] — Participants in this study arm were not provided this treatment, please see Baseline Measure Description. | 10.6 [4 to 21] | 10.6 [4 to 21]

OUTCOME MEASURES:

1. Primary Outcome: Photoactive Porphyrins Level
Description: Photoactive porphyrins levels on the skin surface of acne patients, part 1, measured by in vivo fluorescence spectroscopy
Time Frame: 1.5 hours after cream application
Measure: Mean (95% Confidence Interval); unit: Fluorescence intensity unit
Arm/Group | Part 1: Area Cleaned With Saline and Occluded With Tegaderm | Area Cleaned With Saline | Area Cleaned With Ethyl Alcohol Solution
Number analyzed (Participants) | 12 | 12 | 12
Fluorescence intensity unit | 33.0 [24.8 to 41.3] | 24.8 [20.4 to 29.1] | 19.7 [15.2 to 24.1]

2. Primary Outcome: Photoactive Porphyrins Level
Description: as for outcome 1
Time Frame: 3 hours after cream application
Measure: Mean (95% Confidence Interval); unit: Fluorescence intensity unit
Arm/Group | Part 1: Area Cleaned With Saline and Occluded With Tegaderm | Area Cleaned With Saline | Area Cleaned With Ethyl Alcohol Solution
Number analyzed (Participants) | 12 | 12 | 12
Fluorescence intensity unit | 59.3 [45.4 to 73.2] | 38.3 [31.6 to 45.1] | 30.1 [23.2 to 37.0]

3. Primary Outcome: Photoactive Porphyrins Level
Description: Photoactive porphyrins levels on the skin surface of acne patients, part 2, measured by in vivo fluorescence spectroscopy
Time Frame: 3 hours after cream application
Measure: Mean (95% Confidence Interval); unit: Fluorescence intensity unit
Arm/Group | Visonac Wiped Off After 1 Hour | Visonac Left on Skin for 24 Hours in Area 1 | Visonac Left on Skin for 24 Hours in Area 2
Number analyzed (Participants) | 8 | 8 | 8
Fluorescence intensity unit | 35.3 [16.4 to 54.1] | 33.5 [20.4 to 46.6] | 37.3 [21.4 to 53.1]

4. Primary Outcome: Photoactive Porphyrins Level
Description: as for outcome 3
Time Frame: 8 hours after cream application
Measure: Mean (95% Confidence Interval); unit: Fluorescence intensity unit
Arm/Group | Visonac Wiped Off After 1 Hour | Visonac Left on Skin for 24 Hours in Area 1 | Visonac Left on Skin for 24 Hours in Area 2
Number analyzed (Participants) | 8 | 8 | 8
Fluorescence intensity unit | 21.6 [12.4 to 30.8] | 38.2 [23.1 to 53.3] | 44.3 [24.6 to 64.1]

5. Primary Outcome: Photoactive Porphyrins Level
Description: as for outcome 3
Time Frame: 12 hours after cream application
Measure: Mean (95% Confidence Interval); unit: Fluorescence intensity unit
Arm/Group | Visonac Wiped Off After 1 Hour | Visonac Left on Skin for 24 Hours in Area 1 | Visonac Left on Skin for 24 Hours in Area 2
Number analyzed (Participants) | 8 | 8 | 8
Fluorescence intensity unit | 16.8 [11.8 to 21.8] | 33.9 [23.5 to 44.4] | 38.1 [21.8 to 54.5]

6. Primary Outcome: Photoactive Porphyrins Level
Description: as for outcome 3
Time Frame: 24 hours after cream application
Measure: Mean (95% Confidence Interval); unit: Fluorescence intensity unit
Arm/Group | Visonac Wiped Off After 1 Hour | Visonac Left on Skin for 24 Hours in Area 1 | Visonac Left on Skin for 24 Hours in Area 2
Number analyzed (Participants) | 8 | 8 | 8
Fluorescence intensity unit | 13.1 [8.5 to 17.7] | 25.8 [17.0 to 34.6] | 25.9 [17.6 to 34.2]

ADVERSE EVENTS:
Arm/Group | 3 Areas Per Patient, 3 Hours | 3 Areas Per Patient, 24 Hours
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 5/12 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 Areas Per Patient, 3 Hours (N=12) | 3 Areas Per Patient, 24 Hours (N=8)
Itching (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (4)
Increased number of pimples (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Burning (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No